CLINICAL TRIAL: NCT04751994
Title: Enhancing Brain Development by Early Iron Supplementation of African Infants: An Enabling Pilot Study
Brief Title: Iron Babies Pilot Supplementation Trial
Acronym: Iron Babies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LEO 19092
Record Dates: First submitted 2021-01-27; First posted 2021-02-12 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Iron-deficiency; Anaemia in Early Infancy
Keywords: anaemia, infant
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia | interventions — ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Daily iron (7.5mg/day as ferrous sulphate) or placebo drops starting from six to ten weeks of age for 98 days.
  Please note that the daily iron supplement is the intervention product/drug
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a two-arm, randomised, placebo-controlled double-blind study. Children will be randomised (1:1) to iron drops or placebo arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Iron supplement/ ferrous sulphate syrup (Experimental): administration of daily iron drops, 7.5mg/day iron as ferrous sulphate
  Interventions: Dietary Supplement: Iron drops/Ferrous sulphate
- supplement with placebo (Placebo Comparator): administration of daily placebo drops
  Interventions: Dietary Supplement: Placebo drops

INTERVENTIONS:
Dietary Supplement: Iron drops/Ferrous sulphate — participant will consume daily drops of iron
  Other Names: Ferrous Sulphate syrup
  Arms: Iron supplement/ ferrous sulphate syrup
Dietary Supplement: Placebo drops — Participants will consume daily drops of placebo
  Other Names: Sorbitol Solution 70%
  Arms: supplement with placebo

SUMMARY:
2-arm, double blind, placebo controlled, randomised trial, with 50 6-week-old infants per arm randomized to 98 days of daily iron (1.5mg/kg/day as ferrous sulphate) or placebo drops

DETAILED DESCRIPTION:
Healthy infants will be randomised to receive daily supplementation from 6-20wks of either a) iron drops or b) placebo drops. Infants with significant illness or any clinical syndromes that would affect interpretation will be excluded. Low birthweight infants and infants born prematurely will not be excluded. Venous blood samples will be collected at enrollment (age 6 weeks) and after 14 weeks (98 days) of iron/placebo supplementation.

Participants will be visited daily in their villages by Fieldworkers (FW) to administer the iron/placebo dose and will interview mothers to complete a short health questionnaire. The iron will be dosed at 75% of WHO guideline dose (ie 1.5mg/kg/day). Weekly, a more detailed morbidity and breastfeeding questionnaires will be administered. Infants will be weighed and measured monthly, along with a faecal sample being taken.

During the daily visits, the FWs will record any adverse events (AEs) and ensure the safety of participants. If a child is found unwell or if the mother/guardian reports that the child is unwell, the study nurse will check on the child and decide on treatment/referral to the nearest health centre

ELIGIBILITY:
Inclusion Criteria:

* Infants (male or female) from 6 weeks to 10 weeks of age.
* Breast fed infants (with plans to continue breastfeeding through 6 months of age).
* Parent/guardian with participant reside in study site area and are able and willing to adhere to all protocol visits and procedures (willingness to stay in the study area for the 14 weeks of supplementation).
* Healthy with no current illness and no chronic health problems.
* Signed or fingerprinted informed consent obtained from participants parent/guardian

Exclusion Criteria:

* Low birthweight babies (ie less than 2.5kg at birth) or babies born prematurely (ie less than 37 weeks) will NOT be excluded.
* Formula fed infants or those planning to terminate exclusive breast feeding before 6months of age.
* Acute illness (once acute illness is resolved, if appropriate, as per investigator assessment, participant may be re-revaluated for eligibility)
* Fever (for eligibility purpose defined as a body temperature greater than 37.5°C or mother report of fever) within 3 days prior to study initiation (once fever/acute illness is resolved, if appropriate, as per investigator assessment, participant may be re-revaluated for eligibility).
* Administration of any investigational drug within 30 days prior to study initiation or planned administration during the study period.
* Unwilling to avoid (their child to avoid) the ingestion of supplements or herbal/other traditional medications during the study period.
* Any history of or evidence for chronic clinically significant (as per investigator assessment) disorder or disease (including, but not limited to, immunodeficiency, autoimmunity, congenital abnormality, bleeding disorder, and pulmonary, cardiovascular, metabolic, neurologic, renal, or hepatic disease).
* Any history of human immunodeficiency virus, chronic hepatitis B or chronic hepatitis C infections.
* History of meningitis, seizures, Guillain-Barré syndrome, or other neurological disorders.
* Any condition that in the opinion of the investigator might compromise the safety or well- being of the participant or compromise adherence to protocol procedures

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
serum iron level | at day 0 and at day 99
  Serum iron concentration at days 0 and 99

SECONDARY OUTCOMES:
Haemoglobin concentration | at day 0 and at day 99
  Haemoglobin concentration at days 0 and 99
Percentage of infants with anaemia | at day 99
  Percentage of infants with anaemia (defined as: Hb< 110g/L, )
breast feeding | weekly up to week 14
  Duration of breast feeding assessed weekly, up to study day 98.
maternal reported illnesses | daily up to day 99
  Proportion of maternal-reported illnesses assessed daily up to study day 99.
adverse events assessment | daily up to day 99
  Proportion of adverse events assessed daily, up to study day 99
Serious adverse events (SAE) assessment | daily up to day 99
  Proportion of serious adverse events assessed daily, up to study day 99
raised inflammatory markers assessment | after 98 days of supplementation
  Proportion of raised inflammatory markers (CRP/AGP)
iron deficiency anemia (Hb < 11 g/dL & sTfR/logFerritin ratio < 2.0 and ferritin < 12 ug/L or < 30 ug/L in the presence of inflammation | at day 0 and day 99
  Proportion of children that are iron deficiency anaemia (Hb < 11 g/dL & sTfR/logFerritin ratio < 2.0 and ferritin < 12 ug/L or < 30 ug/L in the presence of inflammation)
Fecal iron after supplementation | day 0 and day 99
  Fecal iron assessed at day 0 and day 99
Iron regulation | day 0 and day 99
  Hepcidin levels at day 0 and day 99
Reticulocytes at day 0 and day 99 | day 0 and day 99
  Reticulocytes at day 0 and day 99
Erythropoietin at days 0 and 99 | day 0 and 99
  Erythropoietin at days 0 and 99
Erythroferrone at days 0 and 99 | day 0 and 99
  Erythroferrone at days 0 and 99

CONTACTS AND LOCATIONS:
Overall Officials: Carla Cerami, MD, PhD, Principal Investigator — Medical Research Council The Gambia at London School of Hygiene & Tropical Medicine
Locations (1):
- Keneba Field Station, Keneba, The Gambia

IPD SHARING:
Plan to Share IPD: No
Data will be kept anonymous. There are currently no plans to share individual patient data beyond the investigator team. However, following all requisite approvals, an anonymized copy of the data can be made available for sharing. All key findings from this study will be submitted for publication in peer-reviewed journals.

REFERENCES:
- [Derived] Stelle I, Bah M, Silverio SA, Verhoef H, Comma E, Prentice AM, Moore SE, Cerami C. Iron supplementation of breastfed Gambian infants from 6 weeks to 6 months of age: protocol for a randomised controlled trial. Wellcome Open Res. 2022 Jan 18;7:16. doi: 10.12688/wellcomeopenres.17507.1. eCollection 2022. PMID 36874582